CLINICAL TRIAL: NCT06221527
Title: Assessment of Healing Properties Using Hyaluronic Acid Topical Application in Parasymphyseal Fracture Fixation: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, aisha khaled mansour, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Omfs 3 3 16
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Maxillofacial Trauma
Keywords: parasymphyseal fracture; hyaluronic acid

STUDY DESIGN:
Intervention Model Description: comparison between healing properties using hyaluronic acid topical application and not using it in parasymphyseal fracture
Who Masked: Participant, Outcomes Assessor
Masking Description: Double(Participant, Outcome Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): fixation of parasymphyseal fracture using two four-hole titanium miniplates that will be placed on inferior border and another one on superior border.
  Interventions: Procedure: conventional group
- study group (Active Comparator): placement of hyaluronic acid will be carried over gel foam and placed between fractured segments before plate fixation.
  fixation of parasymphyseal fracture using two four-hole titanium miniplates that will be placed on inferior border and another one on superior border.
  Interventions: Procedure: conventional group

INTERVENTIONS:
Procedure: conventional group — fixation of parasymphyseal fracture using two four-hole titanium miniplates that will be placed on inferior border and another one on superior border
  Other Names: study group,- Placement of hyaluronic acid paste will be carried over gel foam and placed between fractured segments of parasymphysial before plate fixation

SUMMARY:
HA is favorable for osteogenesis, enhancing bone growth, acting a vector for osteoinductive compounds and promoting even distribution and increased density of newly formed bone, thereby altering the scaffold morphology and improving mineralization. In this study 22 volunteers will be included in this study, the volunteers will be randomly distributed into two groups each containing 11 volunteers, one group will be treated by hyaluronic acid before fixation and the other group will be treated by fixation only without placement of hyaluronic acid, to compensate for drop out 13 volunteers per group

DETAILED DESCRIPTION:
Patients of both groups will be subjected to:

1. Clinical assessment including case history including personal data,medical,surgical history and family history
2. Radiographic assessment includes preoperative digital panomora to evaluate fracture and to conclude presence or absence of any foreign body or pathological pathosis.
3. Signing the informed consent will be done after explaining surgical procedure. All the patients will be nasally intubated, scrubbed and draped in the standard manner, followed by intra-oral and extra-oral povidone-iodine (Betadine)swabbing.

Local anesthesia containing vasoconstrictor will be injected in the vestibule Incision at lower anteriors will be done in the mucosa in a curvilinear fashion 10-15mm away from the attached gingiva, the incision distal to the canine will be 5 mm from the attached gingival to be superior to the mental nerve.

Submucosal dissection will be done to expose the mentalis muscle, followed by mucoperiosteal flap elevation till inferior border exposing the fracture line.

The fracture segments will be reduced after curettage and removal of any debris.

MMF will be done to ensure proper occlusion. Two four-hole titanium miniplates will be placed on inferior border and another one on superior border.

For the intervention group: placement of hyaluronic acid paste will be carried over gel foam and placed between fractured segments before plate fixation.

For the control group: no hyaluronic acid paste will be applied during fixation only gel foam between fractures segments without any additives.

Suturing using 4-0 resorbable sutures will take place after MMF release in layers, anteriorly mentalis muscle will be closed first to prevent chin drooping followed by a continuous running closure of mucosa.

Elastic dressing will be applied over chin region supporting the soft tissues and preventing hematoma formation.

Post-operative care:

Avoid traumatization of the surgical site. All patients will be instructed to apply ice packs over submental area for 15 minutes per hour for 24 hours postoperatively.

All patients will be given postoperative medication as follows:

Anti-inflammatory drug diclofenac potassium (Cataflam50mg)2tabletsevery8hoursforaweek to relieve pain Antibiotic drug Amoxicillin/clavulanic acid tablets (Hibiotic 1gm)1gm every 12 hours for 7 days

-Benzethonium Chloride (Antiseptol mouthwash), starting from the day after the surgery 3 times daily for 10 days.

Instruct the patient not to touch or manipulate the surgical area. No consumption of tobacco for one week postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral Para symphyseal fracture
* Systemically healthy patients (American Society of Anesthesiologists -ASA I and II)
* Age of the patient above 16 years to 60 years old
* Patient of both sexes
* Patients willing for the surgical procedure and follow up with an informed consent.

Exclusion Criteria:

* Bad oral hygiene
* smokers (>10cigarettes/day)
* Existence of a bone metabolic disease; currently taking drugs that might influence bone metabolism
* Radiotherapy or chemotherapy form malignancy
* Patients who refused to sign consent form

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction(score) | at one week and three months intervals
  Patient satisfaction survey through score

SECONDARY OUTCOMES:
Fracture gap distance(mm) | immediate postoperative and four months intervals
  Radiographically(CBCT) through millimeter

OTHER OUTCOMES:
BV\TV (Bone Volume Fraction ) (%) | immediate postoperative and four months intervals
  Radiographically(CBCT) through percent (%)
Pain(VAS) | at one week and three months intervals
  Questionnaire through VAS
Wound dehiscence(Binary) | at one week and three months intervals
  Clinically through binary